CLINICAL TRIAL: NCT01349556
Title: Prevention of Epidermal Growth Factor Receptor Inhibitor-Associated Dermatologic Toxicities by Pre-treatment With Topical Tretinoin
Brief Title: Prevention of Drug Rash From Certain Cancer Therapies Using Tretinoin Cream
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to volunteer disinterest in participating.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Anna Chien, Assistant Professor, Co-Director, Cutaneous Translational Research Program, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NA_00042104
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Medication Reaction
Keywords: cancer; chemotherapy; EGFR inhibitors; tretinoin; EGFRi drug rash
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Neoplasms | interventions — Tretinoin

ARMS (1):
- Tretinoin pre-treatment (Experimental)
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Tretinoin — tretinoin 0.025% cream

SUMMARY:
This research is being done to study whether using of topical tretinoin can help prevent the common rash that patients often get while taking epidermal growth factor inhibitor (EGFR-I) medications such ascetuximab or erlotinib.

Patients taking EGFR-I medications often develop skin irritation and acne-like bumps on their face, chest, and other areas. This rash from EGFR-I's is often treated with moisturizers and topical or oral antibiotics. However, there has not yet been a study looking at a way to prevent this common side effect from occurring, and topical tretinoin may be useful in reducing the rash.

Tretinoin 0.025% cream is approved by the Food and Drug Administration (FDA) for the treatment of acne, acne scarring, and photodamage. It is not approved for use in preventing rashes associated with EGFR-I's.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Scheduled to begin treatment with an EGFR inhibitor drug

Exclusion Criteria:

* Pregnant or nursing
* History of bleeding disorder
* History of keloids or large, thick, puffy-looking scars in the last 10 years
* Used topical retinoids in the last year (e.g. tretinoin/Retin-A, adapalene/Differin, tazarotene/Tazorac)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
EGFRi rash severity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna L Chien, MD, Principal Investigator — Johns Hopkins Dermatology